CLINICAL TRIAL: NCT02789449
Title: Non-invasive Estimation of Pulmonary Capillary Blood Volume in Pre- and Postcapillary Pulmonary Hypertension - a Pilot Study
Brief Title: Estimation of Pulmonary Capillary Blood Volume in Pre- and Postcapillary Pulmonary Hypertension
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: 27-203 ex 14-15
Record Dates: First submitted 2016-04-22; First posted 2016-06-03 (Estimated); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Hypertension Pulmonary
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- precapillary: patients with PH and PAWP<12mmHg
  Interventions: Other: assessment of DLNO and DLCO
- postcapillary: patients with PH and PAWP>18mmHg
  Interventions: Other: assessment of DLNO and DLCO

INTERVENTIONS:
Other: assessment of DLNO and DLCO

SUMMARY:
The aim of the study is to investigate the role of the non-invasive assessment of nitric oxyde (NO) diffusion capacity (DLNO) in the differential diagnosis of different forms of pulmonary hypertension (PH). DLNO alone and in combination with the measurement of carbon monoxide (CO) diffusion capacity (DLCO) may help to differentiate between pre- and postcapillary forms of pulmonary hypertension. This hypothesis is based on the fact that NO has a much higher affinity to hemoglobin as compared to CO and may therefore its decrease may more specifically identify the limiting factors between the alveolar space and the lung capillaries including left heart failure (cardiac edema).

As there are no available published data yet to answer this question investigators aim to perform a small pilot study. The results of this study may allow the planning of a prospective study.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing right heart catheterization
* patients with clear precapillary PH (PAWP<12mmHg) or clear postcapillary PH (PAWP>18mmHg)
* signed informed consent

Exclusion Criteria:

* patients unable to perform the DLCO test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with PH
Sampling Method: Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2015-11; Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Difference in DLNO (in mmol/min/kPa) between the two predefined groups (patients with clear precapillary PH (PAWP<12mmHg) vs. clear postcapillary PH (PAWP>18mmHg)) | one hour

CONTACTS AND LOCATIONS:
Overall Officials: Horst Olschewski, MD, Principal Investigator — Medical University of Graz
Locations (1):
- Medical University Graz, Division of Pulmonology, Graz, Styria, Austria

IPD SHARING:
Plan to Share IPD: No